CLINICAL TRIAL: NCT02564627
Title: Percutaneous Electrical Neurostimulation (PENS) of Dermatome T6 With an Ambulatory Self-applied Patch vs PENS of Dermatome T6 With Conventional Procedure: Effect on Appetite and Weight Loss in Moderately Obese Patients
Brief Title: PENS T6 With Ambulatory Self-applied Patch vs Conventional Procedure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abdel Kadar Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KC15-02
Record Dates: First submitted 2015-09-25; First posted 2015-10-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Self-applied patch (Experimental): The patients will use a self-applied patch weekly for PENS of dermatome T6. A 1200 Kcal/day diet will be also prescribed.
  Interventions: Procedure: Self-applied patch; Dietary Supplement: 1200 Kcal/day diet
- Conventional procedure (Active Comparator): The patient will attend weekly the Outpatient Clinic for receiving the PENS of dermatome T6. The procedure will be performed by the Medicine Doctor. A 1200 Kcal/day diet will be also prescribed.
  Interventions: Procedure: Conventional procedure; Dietary Supplement: 1200 Kcal/day diet
- 1200 Kcal/day diet (Other): A 1200 Kcal/day diet will be also prescribed.
  Interventions: Dietary Supplement: 1200 Kcal/day diet

INTERVENTIONS:
Procedure: Self-applied patch — An ambulatory self-applied patch will be placed weekly by the patients for PENS of dermatome T6.
  Arms: Self-applied patch
Procedure: Conventional procedure — PENS of dermatome T6 will be applied by the MD in the Outpatient Clinic.
  Arms: Conventional procedure
Dietary Supplement: 1200 Kcal/day diet — A 1200 Kcal/day diet will be prescribed.

SUMMARY:
A prospective randomized study, including moderately obese patients will be included. Patients will be randomized in 3 groups:

* PENS of dermatome T6 with an ambulatory self-applied patch + 1200Kcal/day diet
* PENS of dermatome T6 with conventional procedure + 1200Kcal/day diet
* Only 1200Kcal/day diet

The effect on appetite and weight loss will be investigated.

DETAILED DESCRIPTION:
A prospective randomized study, including moderately obese (BMI 30-39 Kg/m2) patients will be included. Patients will be randomized in 3 groups:

* PENS of dermatome T6 with an ambulatory self-applied patch + 1200Kcal/day diet
* PENS of dermatome T6 with conventional procedure (weekly stimulation in the Outpatient Clinic) + 1200Kcal/day diet
* Only 1200Kcal/day diet

The effect on appetite and weight loss will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Moderately obese patients (BMI 30-39 kg/m2)

Exclusion Criteria:

* Endocrinological diseases causing obesity
* Heart pacemaker
* Previous bariatric procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Appetite will be quantified with a visual analogic scale | 12 weeks
  Appetite will be quantified weekly during the 12 weeks of treatment. Appetite will be quantified with a visual analogic scale (0= absence of appetite, 10=uncontrollable appetite)

SECONDARY OUTCOMES:
Weight loss | 12 weeks
  Appetite will be quantified weekly during the 12 weeks of treatment
Compliance will be evaluated by means of a food diary filled by the patients and evaluated by a nutritionist | 12 weeks
  The compliance with the 3 arms of treatment will be investigated. Diet complience will be evaluated by means of a food diary filled by the patients and evaluated by a nutritionist.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Abdel Kadar, Principal Investigator — Kadar Clinic

REFERENCES:
- [Derived] Abdel-Kadar M. Percutaneous Electrical Neurostimulation (PENS) of Dermatome T6 with an Ambulatory Self-applied Patch vs PENS of Dermatome T6 with Conventional Procedure: Effect on Appetite and Weight Loss in Moderately Obese Patients. Obes Surg. 2016 Dec;26(12):2899-2905. doi: 10.1007/s11695-016-2214-0. PMID 27289457